CLINICAL TRIAL: NCT00313625
Title: A Phase II Study of Intravenous Melphalan and Busulfan Followed by HLA-Matched, Allogeneic Peripheral Blood Stem Cell Transplant for the Treatment of Multiple Myeloma
Brief Title: Melphalan and Busulfan Followed By Donor Peripheral Stem Cell Transplant, Tacrolimus, and Methotrexate in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: William I. Bensinger, Fred Hutchinson Cancer Research Center
Masking: None | Purpose: Treatment
Other Study IDs: 2018.00; FHCRC-2018.00; CDR0000467231 (Registry Identifier: PDQ)
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Busulfan; Melphalan; Methotrexate; Tacrolimus; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: busulfan
Drug: melphalan
Drug: methotrexate
Drug: tacrolimus
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy, such as melphalan and busulfan, before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving tacrolimus and methotrexate before or after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving melphalan together with busulfan followed by donor peripheral stem cell transplant, tacrolimus, and methotrexate works in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate transplant-related mortality in patients with multiple myeloma treated with a myeloablative conditioning regimen comprising melphalan and busulfan followed by HLA-matched, allogeneic peripheral blood stem cell transplantation (PBSCT) and graft-vs-host disease prophylaxis with tacrolimus and methotrexate.

Secondary

* Determine the disease response in patients treated with this regimen.
* Determine the 1-year progression-free survival and overall survival in patients treated with this regimen.

OUTLINE:

* Conditioning regimen: Patients receive melphalan IV over 30 minutes on day -6 and busulfan IV over 3 hours on days -5 to -3.
* Peripheral blood stem cell transplantation (PBSCT): Patients undergo HLA-matched, related donor, allogeneic PBSCT on day 0.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive tacrolimus IV continuously or orally twice daily beginning on day -2 and continuing until day 80 followed by a taper until day 180 in the absence of GVHD or disease progression. Patients also receive methotrexate IV on days 1, 3, 6, and 11.

After completion of study treatment, patients are followed every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma

  * Stage I disease with disease progression during the second of ≥ 2 lines of prior therapy
  * Stage II or III disease, meeting 1 of the following criteria:

    * Failed to achieve at least a partial response after ≥ 2 courses of prior therapy
    * Progressive disease after ≥ 2 courses of prior therapy
    * Presented with high-risk features at diagnosis, including any of the following:

      * Cytogenetic abnormality
      * Del 13 or 4,14 by fluorescent in situ hybridization (FISH)
      * Elevated lactic dehydrogenase
      * Beta 2 microglobulin > 5.5
      * Circulating peripheral blood plasma cells
  * Any stage disease with disease progression > 6 months after prior autologous stem cell transplantation
* Availability of an HLA-matched, related donor between 12 and 75 years of age*

  * No bone marrow donors NOTE: *Donors > 75 years of age are eligible at the discretion of the principal investigator

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Creatinine clearance > 60 mL/min
* Bilirubin ≤ 2.5 mg/dL
* ALT/AST < 2 times upper limit of normal
* Cardiac ejection fraction ≥ 49%
* DLCO ≥ 50% corrected
* FEV_1 ≥ 60%
* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No cirrhosis
* No chronic inflammatory or fibrotic liver disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 6 months since prior autologous transplantation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Transplant-related mortality at 180 days

SECONDARY OUTCOMES:
Disease response (complete response)
Progression-free survival
Overall survival at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: William I. Bensinger, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States